CLINICAL TRIAL: NCT03045939
Title: Cervical Ripening With the Double Balloon Device for 6 Hours Compared With 12 Hours. A Randomized Multicenter Controlled Trial
Brief Title: Cervical Ripening With the Double Balloon Device for 6 Hours Compared With 12 Hours
Acronym: DoubleCRIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Inna.bleicher, principle investigator Dr. Inna Bleicher, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BNZ-0115-16
Record Dates: First submitted 2017-01-24; First posted 2017-02-08 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Induction of Labor; Unfavorable Cervix
Keywords: cervical ripening; labor induction; double balloon device; cervical ripening device; unfavorable cervix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 hours (Other): This arm is the standard management that includes insertion of the DBD into the cervical canal according to manufacture guidelines, removal after 12 hours followed by artificial rupture of membranes and oxytocin infusion according to departments protocol. (a total of 10 units of oxytocin is infused, initiated with 10 cc/h, increased by 10cc every 20-30 min until 3-5 contractions are present, total of not more than 120 cc\h)
  Interventions: Device: cervical ripening device
- 6 hours (Active Comparator): Removal of the DBD after 6 hours, followed by artificial rupture of membranes and oxytocin infusion according to departments protocol. (a total of 10 units of oxytocin is infused, initiated with 10 cc/h, increased by 10cc every 20-30 min until 3-5 contractions are present, total of not more than 120 cc\h)
  Interventions: Device: cervical ripening device

INTERVENTIONS:
Device: cervical ripening device — insertion of the double balloon device for 12 hours (standard care) vs 6 hours, following oxytocin IV infusion according local protocol guidelines as mentioned above
  Other Names: atad double balloon device

SUMMARY:
This study will evaluate the insertion of double balloon device (DBD) for cervical ripening for 12 h vs 6 hours.

DETAILED DESCRIPTION:
This randomized controlled study is designed to:

1. To assess and compare the Bishop score when removing the DBD 12 hours' vs 6hours' after insertion.
2. To compare the efficacy (vaginal delivery rate and time to VD) in the two arm groups

200 women are expected to be randomized in to two arms. One will be randomized to DBD removal after 12 hours and the other to DBD removal after 6 hours.

Each patient will sign an informed consent.

The following screening will be completed: medical and gynecological history, general physical and gynecological examination, ultrasonography to exclude contraindication to vaginal delivery or insertion if the DBD and non stress test (NST) for baseline. Bishop score will be assessed.

After confirming eligibility for study, randomization into the following groups will take place.

Insertion of the DBD and removal 6 hours following its insertion. Insertion of the DBD and removal 12 hours following its insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Parous patients 18 years of age or older.
2. Diagnosed to be parous pregnant women with an indication for induction of labour.
3. Having a Bishop score of 5 or less.
4. Diagnosed as having a singleton pregnancy in a vertex presentation, with intact membranes, and no significant regular uterine contraction at gestational age of 37 completed gestational weeks or more.
5. Willingness to comply with the protocol for the duration of the study.
6. Have signed the informed consent.

   -

Exclusion Criteria:

1. A non -vertex presentation
2. Placenta previa
3. Ruptured membranes
4. Documented labour
5. Foetal distress necessitating immediate intervention
6. Proven malignancy of the cervix
7. Active inflammatory or purulent condition of the lower genital tract
8. Twin pregnancy
9. Any other contraindication for vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
time from insertion of the DBD to delivery | minutes or hours from insertion to delivery, assessed up to an estimated total of 24 hours
  the time from insertion of the DBD until delivery will be assessed for each patient from each arm by hours/minutes

SECONDARY OUTCOMES:
rate of vaginal delivery | 1 year
  calculation of the rate of vaginal delivery in each arm will be calculated by number of Vaginal deliveries in each arm and the percentage.
maternal and neonatal adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Mc, Haifa, Israel

REFERENCES:
- [Derived] Sammour R, Dikopoltsev E, Sagi S, Vitner D, Bleicher I. Cervical ripening with a double balloon device for 6 h in patients with a long cervix: Secondary analysis of a randomized controlled trial. Int J Gynaecol Obstet. 2025 Mar;168(3):1055-1059. doi: 10.1002/ijgo.15955. Epub 2024 Oct 24. PMID 39445570
- [Derived] Bleicher I, Dikopoltsev E, Kadour-Ferro E, Sammour R, Gonen R, Sagi S, Eshel A, Nussam L, Vitner D. Double-Balloon Device for 6 Compared With 12 Hours for Cervical Ripening: A Randomized Controlled Trial. Obstet Gynecol. 2020 May;135(5):1153-1160. doi: 10.1097/AOG.0000000000003804. PMID 32282603